CLINICAL TRIAL: NCT03680690
Title: Pregnancy Rate in Women With Normal Uterine Cavity and Those With Corrected Uterine Lesions in ICSI Cycles
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Momen Ahmed Mohammed Kamel, Principle investigator, Assiut University
Other Study IDs: pregnancy rate in ICSI cycles
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Intracytoplasmic Sperm Injection
MeSH Terms: interventions — Hysteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: women with normal uterus,detected by hysteroscopy.
  Interventions: Procedure: hysteroscopy
- Group B: Women with detected or corrected uterine cavitary lesions by hysteroscopy.
  Interventions: Procedure: hysteroscopy

INTERVENTIONS:
Procedure: hysteroscopy — office hysteroscopy will be done for all candidates and operative correction of detected lesions will be carried on.
  Other Names: hysteroscopic uterine lesion detection or correction

SUMMARY:
The aim of the current study is to investigate the pregnancy rate in women with normal uterine cavity and those detected or corrected uterine cavitary lesions, assessed by hysteroscopy in ICSI cycles.

DETAILED DESCRIPTION:
Intrauterine pathology has been reported in up to 25% of infertile women having IVF treatment and in as many as 50% of women with recurrent implantation failure, leading to suggestions that correction of such pathology could improve treatment outcome. Hysteroscopy allows visual assessment of the cervical canal and uterine cavity and provides the opportunity to operate in the same setting. Routine outpatient hysteroscopy before starting IVF has been postulated to diagnose and treat abnormalities of the cervix and uterine cavity and hence improve IVF outcome.

A systematic review of published studies suggested that outpatient hysteroscopy in the menstrual cycle preceding an IVF treatment cycle could significantly increase the clinical pregnancy rate in women who had previously had recurrent implantation failure, even when no hysteroscopic abnormality was detected.

However, the result of the TROPHY study - published in the Lancet in 2016 concluded that Outpatient hysteroscopy before IVF in women with a normal ultrasound of the uterine cavity and a history of unsuccessful IVF treatment cycles does not improve the livebirth rate and they recommended that further research into the effectiveness of surgical correction of specific uterine cavity abnormalities before IVF is warranted.

An MD thesis done in our department on the evaluation of the endometrial cavity in infertile patients and prior to IVF recommended that there is an urgent need to RCT to emphasize the benefit of removal of the detected intrauterine lesions before proceeding to IVF.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 38 years old.
* An indication for IVF/ICSI.
* Normal 2D transvaginal U/S assessment of the uterine cavity, or abnormal cavity detected by 2D ,3D and HSG.
* Women with primary or secondary infertility.
* Women with BMI between 20 & 35.

Exclusion Criteria:

* Refusal to join the study.
* Untreated tubal hydrosalpinges.
* Poor responders as assessed by AFC 4 or less ,AMH O.8 ng/dl (nice 2013).

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — infertile females
Study Population: all infertile females will be assesed in IVF unite of women's health Hospital and will be recruted according to the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7th week of pregnancy for cardiac pulsations.
  Clinical pregnancy rate Will be evaluated

SECONDARY OUTCOMES:
Chemical pregnancy rate Chemical pregnancy rate | 4 weeks
  Chemical pregnancy rate
  Chemical pregnancy rate
Implantation rate | 6 weeks
  Implantation rate for assessment of implanted embryos
Abortion rate | up to 28 week
  Abortion rate will be observed
Preterm labour rate | 9 months
  Delivary before term 37 weeks of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Youssef, MD/MSC, Study Chair — women's health hospital,Assiut university; Ibrahim Mohammed, MD/MSc, Study Director — women's health hospital,Assiut university; Sayed Moustafa, MD/MSC, Principal Investigator — women's health hospital,Assiut university; Ahmed Kamel, MSC/MBBh, Principal Investigator — women's health hospital,Assiut university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Polanski LT, Baumgarten MN, Quenby S, Brosens J, Campbell BK, Raine-Fenning NJ. What exactly do we mean by 'recurrent implantation failure'? A systematic review and opinion. Reprod Biomed Online. 2014 Apr;28(4):409-23. doi: 10.1016/j.rbmo.2013.12.006. Epub 2014 Jan 17. PMID 24581986
- [Result] Coughlan C, Walters S, Ledger W, Li TC. A comparison of psychological stress among women with and without reproductive failure. Int J Gynaecol Obstet. 2014 Feb;124(2):143-7. doi: 10.1016/j.ijgo.2013.08.006. Epub 2013 Oct 31. PMID 24290538
- [Result] Zeyneloglu HB, Onalan G. Remedies for recurrent implantation failure. Semin Reprod Med. 2014 Jul;32(4):297-305. doi: 10.1055/s-0034-1375182. Epub 2014 Jun 11. PMID 24919029
- [Result] Papathanasiou A, Bhattacharya S. Prognostic factors for IVF success: diagnostic testing and evidence-based interventions. Semin Reprod Med. 2015 Mar;33(2):65-76. doi: 10.1055/s-0035-1545364. Epub 2015 Mar 3. PMID 25734344
- [Result] Moini A, Kiani K, Ghaffari F, Hosseini F. Hysteroscopic findings in patients with a history of two implantation failures following in vitro fertilization. Int J Fertil Steril. 2012 Apr;6(1):27-30. Epub 2012 Jun 19. PMID 25505508
- [Result] Cenksoy P, Ficicioglu C, Yildirim G, Yesiladali M. Hysteroscopic findings in women with recurrent IVF failures and the effect of correction of hysteroscopic findings on subsequent pregnancy rates. Arch Gynecol Obstet. 2013 Feb;287(2):357-60. doi: 10.1007/s00404-012-2627-5. Epub 2012 Nov 27. PMID 23183783
- [Result] Dicker D, Ashkenazi J, Feldberg D, Farhi J, Shalev J, Ben-Rafael Z. The value of repeat hysteroscopic evaluation in patients with failed in vitro fertilization transfer cycles. Fertil Steril. 1992 Oct;58(4):833-5. doi: 10.1016/s0015-0282(16)55338-2. PMID 1426335
- [Result] La Sala GB, Montanari R, Dessanti L, Cigarini C, Sartori F. The role of diagnostic hysteroscopy and endometrial biopsy in assisted reproductive technologies. Fertil Steril. 1998 Aug;70(2):378-80. doi: 10.1016/s0015-0282(98)00147-2. PMID 9696242
- [Result] Levi Setti PE, Colombo GV, Savasi V, Bulletti C, Albani E, Ferrazzi E. Implantation failure in assisted reproduction technology and a critical approach to treatment. Ann N Y Acad Sci. 2004 Dec;1034:184-99. doi: 10.1196/annals.1335.021. PMID 15731311
- [Result] El-Toukhy T, Campo R, Khalaf Y, Tabanelli C, Gianaroli L, Gordts SS, Gordts S, Mestdagh G, Mardesic T, Voboril J, Marchino GL, Benedetto C, Al-Shawaf T, Sabatini L, Seed PT, Gergolet M, Grimbizis G, Harb H, Coomarasamy A. Hysteroscopy in recurrent in-vitro fertilisation failure (TROPHY): a multicentre, randomised controlled trial. Lancet. 2016 Jun 25;387(10038):2614-2621. doi: 10.1016/S0140-6736(16)00258-0. Epub 2016 Apr 27. PMID 27132053